CLINICAL TRIAL: NCT07102537
Title: A Single-Arm, Before- After Clinical Study to Evaluate the Safety and Efficacy of Intella Dermal Filler (Produced by Espad Pharmed Darou Co.) for Correction of Moderate to Severe Nasolabial Folds
Brief Title: Evaluation of Efficacy and Safety of Intella Dermal Filler in Moderate to Severe Nasolabial Folds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Espad Pharmed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INT.ESP.AF.IV.02
Record Dates: First submitted 2025-07-13; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-06

CONDITIONS: Nasolabial Fold Correction
Keywords: nasolabial fold; hyaluronic acid; calcium hydroxyapatite

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intella (hyaluronic acid combined with calcium hydroxyapatite, produced by Espad Pharmed Co.) (Experimental): The injection volume is 1-2 milliliters, determined based on the patient's needs and the injecting physician's discretion. The injection method may be linear or consist of multiple point injections using a 27-gauge needle or a 25-gauge cannula, depending on the physician's preference. During injection, the site and technique are carefully monitored to ensure that the filler is not injected into a blood vessel. If higher volumes are needed, multiple layers may be injected, with each layer positioned perpendicularly over the previous one (cross-hatching technique). After the injection, the area is gently massaged to ensure the volume is harmonized with the surrounding tissue. Immediately after injection, an ice pack is applied to the site for 15 minutes. Two weeks after the initial injection, if corrective injection is needed, an additional session with a maximum of 1 milliliter of filler may be performed.
  Interventions: Device: Hyaluronic acid combined with calcium hydroxyapatite injection

INTERVENTIONS:
Device: Hyaluronic acid combined with calcium hydroxyapatite injection — The filler was injected in nasolabial folds in a before-after setting

SUMMARY:
This single-arm, before-and-after clinical trial evaluated the safety and efficacy of Intella, a combined CaHA and HA dermal filler manufactured by Espad Pharmed Darou Co., for the correction of moderate to severe nasolabial folds. The study involved 30 female participants with a mean age of 48.8 years (range 34-64 years).

After obtaining written informed consent and confirming eligibility criteria, 1 to 2 ml of Intela filler was injected subcutaneously into the bilateral nasolabial fold areas by a dermatologist. Assessments were performed immediately before, immediately after, and at 1, 3, and 6 months post-injection. Evaluation methods included standardized photography, independent physician scoring of wrinkle severity, and measurement of wrinkle volume, depth, and surface area using the VisioFace device. Additionally, ultrasonographic parameters and skin elasticity (R0, R2, R5) were recorded at baseline and follow-up visits. Patient satisfaction and adverse events were also documented during follow-up.

At months 1, 3, and 6, 62.9%, 82.7%, and 73% of participants respectively demonstrated at least a one-grade improvement in wrinkle severity. Also, results showed a statistically significant reduction in nasolabial fold severity at all post-treatment visits (p < 0.01). Significant decreases in wrinkle volume and surface area were observed bilaterally. Skin elasticity (R0) improved significantly at months 3 and 6. The median pain score during injection was low (2/10), with a maximum reported pain of 5/10. Four mild adverse events (swelling, bruising, gel accumulation) were reported in three participants, consistent with expected side effects of similar products. Patient satisfaction scores remained high throughout follow-up, ranging from 7 to 10 out of 10.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have moderate to severe nasolabial folds based on the Allergan scale.
* Participants must be able to comply with the visit schedule and study procedures.
* Participants must have signed the informed consent form and agreed to the 6-month follow-up

Exclusion Criteria:

* History of type 1 hypersensitivity reactions or anaphylaxis.
* Previous allergy or sensitivity to filler components or lidocaine.
* History of hypertrophic or keloid scar formation or bleeding disorders in the nasolabial area.
* Presence of active inflammatory processes, infection, or lesions (malignant/non-malignant) in the nasolabial area.
* History of autoimmune diseases/immunodeficiency or use of immunosuppressive drugs within 6 months prior to or during the study.
* Use of antiplatelet drugs within 72 hours prior to treatment and anticoagulants within 2 weeks prior to or during treatment.
* Pregnancy, breastfeeding, or planning pregnancy in the near future during the study.
* Use of cosmetic treatments in recent months or plans to undergo such treatments in the near future during the study, including:

  1. Botulinum toxin type A injections below the zygomatic arch within 6 months prior to study entry.
  2. Non-permanent dermal filler injections (e.g., bovine collagen, hyaluronic acid) in facial areas within 1 year prior to study entry.
  3. Use of calcium hydroxyapatite, poly-L-lactic acid, or permanent fillers (e.g., silicone) in facial areas at any time before or during the study.
  4. Deep skin peeling procedures such as chemical peeling, laser, dermabrasion, radio frequency within 6 months prior to study entry.
  5. Superficial skin peeling within 6 weeks prior to study entry.
* Other reasons that, according to the investigator's judgment, make the patient unsuitable for study participation (e.g., uncertainty about patient cooperation).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-02-14 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
The number of individuals with at least a one-grade reduction in the severity of both nasolabial folds compared to baseline based on the Allergan scale | Baseline, Week 4
  The scale is from 0 to 4, 0 indicating no wrinkle, and 4 indicating very deep wrinkle, redundant fold (overlapping skin)

SECONDARY OUTCOMES:
The number of individuals with at least a one-grade reduction in the severity of both nasolabial folds compared to baseline based on the Allergan scale | Baseline, Week 12, Week 24
  The scale is from 0 to 4, 0 indicating no wrinkle, and 4 indicating very deep wrinkle, redundant fold (overlapping skin)
Assessment of changes in depth of the right and left nasolabial folds | Baseline, Week 4, Week 12, Week 24
Assessment of changes in surface area of the right and left nasolabial folds | Baseline, Week 4, Week 12, Week 24
Assessment of changes in volume of the right and left nasolabial folds | Baseline, Week 4, Week 12, Week 24
Assessment of changes in dermal thickness in the right nasolabial fold area compared to baseline | Baseline, Week 4, Week 24
Assessment of changes in density in the right nasolabial fold area compared to baseline | Baseline, Week 4, Week 24
Assessment of changes in skin elasticity parameter (R0) in the middle of the right nasolabial fold compared to baseline. | Baseline, Week 12, Week 24
Assessment of changes in skin elasticity parameter (R2) in the middle of the right nasolabial fold compared to baseline. | Baseline, Week 12, Week 24
Assessment of changes in skin elasticity parameter (R5) in the middle of the right nasolabial fold compared to baseline. | Baseline, Week 12, Week 24
Assessment of changes in nasolabial fold severity compared to baseline by GAIS score, using before and after photographs | Baseline, Week 4, Week 12, Week 24
  The scale is from 1 to 5, 1 indicating exceptional improvement i.e., excellent corrective result, and 5 indicating worsened patient i.e., the appearance has worsened compared with the original condition
Consumer satisfaction measured using the Visual Analogue Scale (VAS) (from 0 to 10, where 10 indicates complete satisfaction and 0 indicates complete dissatisfaction) | Day 1, Week 2, Week 4, Week 12, Week 24
Pain intensity assessment using the VAS from 0 to 10 | Day 1, Week 2 (based on physician's assessment regarding the need for a touch-up injection)
  Visual Analogue Scale (VAS): pain intensity scale where 0 indicates no pain and 10 indicates the maximum pain imaginable.
Safety assessment by evaluation of adverse events (AEs) | Day 1, Week 2, Week 4, Week 12, Week 24
  Adverse events (AEs) were assessed at all visits. The severity, seriousness, and causality of each AE were evaluated. The seriousness of AEs was determined according to International Council for Harmonization (ICH-E2B) guidelines, causality was assessed based on World Health Organization (WHO) criteria, and severity was classified as mild, moderate, or severe.

CONTACTS AND LOCATIONS:
Locations (1):
- Orchid Pharmed, Medical Department, Tehran, Tehran Province, Iran

IPD SHARING:
Plan to Share IPD: No
Data produced in the present study are available upon reasonable request from the investigators.